CLINICAL TRIAL: NCT06864143
Title: A Phase 2, Randomized, Observer-blind, Active-control Study to Evaluate the Immunogenicity, Reactogenicity, and Safety of mRNA-1083 (Influenza and COVID-19) Vaccine in Adults ≥18 to <65 Years of Age
Brief Title: A Study to Investigate the Immunogenicity, Reactogenicity, and Safety of mRNA-1083 (Influenza and COVID-19) Vaccine in Adults ≥18 to <65 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1083-P202
Record Dates: First submitted 2025-03-05; First posted 2025-03-07 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Influenza; SARS-CoV-2
Keywords: Influenza; SARS-CoV-2; mRNA-1083; COVID-19; Messenger RNA; Moderna
MeSH Terms: conditions — Influenza, Human; COVID-19 | interventions — Influenza Vaccines; COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- mRNA-1083 Composition 1 Dose A Lot A (Experimental): Participants will receive single intramuscular (IM) injection of mRNA-1083 Composition 1 at Dose Level A Lot A on Day 1.
  Interventions: Biological: mRNA-1083 Composition 1 Dose A Lot A
- mRNA-1083 Composition 1 Dose A Lot B (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 1 at Dose Level A Lot B on Day 1.
  Interventions: Biological: mRNA-1083 Composition 1 Dose A Lot B
- mRNA-1083 Composition 1 Dose B (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 1 at Dose Level B on Day 1.
  Interventions: Biological: mRNA-1083 Composition 1 Dose B
- mRNA-1083 Composition 1 Dose C (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 1 at Dose Level C on Day 1.
  Interventions: Biological: mRNA-1083 Composition 1 Dose C
- mRNA-1083 Composition 2 Dose A (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 2 at Dose Level A on Day 1.
  Interventions: Biological: mRNA-1083 Composition 2 Dose A
- mRNA-1083 Composition 2 Dose B (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 2 at Dose Level B on Day 1.
  Interventions: Biological: mRNA-1083 Composition 2 Dose B
- mRNA-1083 Composition 3 Dose A (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 3 at Dose Level A on Day 1.
  Interventions: Biological: mRNA-1083 Composition 3 Dose A
- mRNA-1083 Composition 3 Dose B (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 3 at Dose Level B on Day 1.
  Interventions: Biological: mRNA-1083 Composition 3 Dose B
- Influenza Vaccine (Active Comparator): Participants will receive single IM injection of Influenza Vaccine on Day 1.
  Interventions: Biological: Influenza Vaccine
- COVID-19 Vaccine (Active Comparator): Participants will receive single IM injection of COVID-19 Vaccine on Day 1.
  Interventions: Biological: COVID-19 Vaccine
- Investigational Influenza Vaccine (Active Comparator): Participants will receive single IM injection of Investigational Influenza Vaccine on Day 1.
  Interventions: Biological: Investigational Influenza Vaccine
- Investigational COVID-19 Vaccine Lot A (Active Comparator): Participants will receive single IM injection of Investigational COVID-19 Vaccine Lot A on Day 1.
  Interventions: Biological: Investigational COVID-19 Vaccine Lot A
- Investigational COVID-19 Vaccine Lot B (Active Comparator): Participants will receive single IM injection of Investigational COVID-19 Vaccine Lot B on Day 1.
  Interventions: Biological: Investigational COVID-19 Vaccine Lot B

INTERVENTIONS:
Biological: mRNA-1083 Composition 1 Dose A Lot A — Sterile liquid for injection
  Arms: mRNA-1083 Composition 1 Dose A Lot A
Biological: mRNA-1083 Composition 1 Dose A Lot B — Sterile liquid for injection
  Arms: mRNA-1083 Composition 1 Dose A Lot B
Biological: mRNA-1083 Composition 1 Dose B — Sterile liquid for injection
  Arms: mRNA-1083 Composition 1 Dose B
Biological: mRNA-1083 Composition 1 Dose C — Sterile liquid for injection
  Arms: mRNA-1083 Composition 1 Dose C
Biological: mRNA-1083 Composition 2 Dose A — Sterile liquid for injection
  Arms: mRNA-1083 Composition 2 Dose A
Biological: mRNA-1083 Composition 2 Dose B — Sterile liquid for injection
  Arms: mRNA-1083 Composition 2 Dose B
Biological: mRNA-1083 Composition 3 Dose A — Sterile liquid for injection
  Arms: mRNA-1083 Composition 3 Dose A
Biological: mRNA-1083 Composition 3 Dose B — Sterile liquid for injection
  Arms: mRNA-1083 Composition 3 Dose B
Biological: Influenza Vaccine — Sterile liquid for injection
  Arms: Influenza Vaccine
Biological: COVID-19 Vaccine — Sterile liquid for injection
  Arms: COVID-19 Vaccine
Biological: Investigational Influenza Vaccine — Sterile liquid for injection
  Arms: Investigational Influenza Vaccine
Biological: Investigational COVID-19 Vaccine Lot A — Sterile liquid for injection
  Arms: Investigational COVID-19 Vaccine Lot A
Biological: Investigational COVID-19 Vaccine Lot B — Sterile liquid for injection
  Arms: Investigational COVID-19 Vaccine Lot B

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, reactogenicity, and safety, of mRNA-1083 multicomponent influenza and COVID-19 vaccine in adults ≥18 to <65 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable.
* Participants who could become pregnant: negative pregnancy test and contraception for at least 28 days prior to Day 1 and for at least 90 days after the study intervention administration.
* Have received ≥2 coronavirus disease 2019 (COVID-19) vaccines, with the last COVID-19 vaccine administered >150 days prior to Day 1.

Exclusion Criteria:

* History of a diagnosis or condition that is clinically unstable or may affect participant safety, assessment of study endpoints, assessment of immune response, or adherence to study procedures.
* Tested positive for influenza by local health authority-approved testing methods within 150 days prior to Day 1.
* History of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 150 days prior to Day 1.
* Received systemic immunosuppressive treatment, including long-acting biological therapies that affect immune responses (eg, infliximab), within 180 days prior to Day 1 or plans to do so during the study.
* Received or plans to receive any vaccine authorized or approved by a local health agency within 28 days prior to Day 1 or plans to do so within 28 days post study injection.
* Received a licensed seasonal influenza vaccine within 150 days prior to Day 1.
* Received a licensed/authorized COVID-19 vaccine within 150 days prior to Day 1.
* Received any investigational influenza vaccine, investigational COVID-19 vaccine, or investigational combination vaccine for influenza and COVID-19 within 12 months prior to Day 1.
* Participated in a clinical study with investigational treatment within 90 days prior to Day 1 (Baseline).

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1320 (Actual)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) as Measured by Hemagglutination Inhibition (HAI) Assay for Influenza | Day 29
Geometric Mean Concentration (GMC) as Measured by Pseudovirus Neutralization Assay (PsVNA) for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) | Day 29
Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs) | Day 1 through 7 days after study injection
Number of Participants With Unsolicited Adverse Events (AEs) | Day 1 through 28 days after study injection
Number of Participants With Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs), Serious Adverse Events (SAEs), and AEs Leading to Discontinuation From the Study | Day 1 through Day 181

SECONDARY OUTCOMES:
Geometric Mean Fold-Rise (GMFR) of Antibodies for Influenza as Measured by HAI Assay | Baseline (Day 1), Day 29
GMFR of Antibodies for SARS-CoV-2 as Measured by PsVNA | Baseline (Day 1), Day 29
Influenza: Percentage of Participants with Seroconversion as Measured by HAI Assay | Baseline (Day 1) to Day 29
  Seroconversion is defined as postinjection level ≥1:40 if baseline is <1:10 or at least a 4-fold rise if baseline is ≥1:10 in HAI antibody titer.
SARS-CoV-2: Percentage of Participants with Seroresponse as Measured by PsVNA | Baseline (Day 1) to Day 29
  Seroresponse is defined as PsVNA concentration change from preinjection baseline below the lower limit of quantification (LLOQ) to postinjection ≥4×LLOQ, or at least a 4-fold rise if baseline is ≥LLOQ.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Headlands Research Scottsdale, Scottsdale, Arizona
  - Artemis Research (Headlands), San Diego, California
  - Clinical Research Atlanta (Headlands), Stockbridge, Georgia
  - Velocity Clinical Research, Boise, Meridian, Idaho
  - DM Clinical Research - Chicago, Melrose Park, Illinois
  - Velocity Clinical Research, Lafayette, Lafayette, Louisiana
  - Velocity Clinical Research, Rockville, Rockville, Maryland
  - DM Clinical Research - Boston, Brookline, Massachusetts
  - DM Clinical Research - Detroit, Southfield, Michigan
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Velocity Clinical Research, Cincinnati, Mt. Auburn, Cincinnati, Ohio
  - Velocity Clinical Research, Cincinnati, Springdale, Cincinnati, Ohio
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Trial Management Associates, LLC, Myrtle Beach, South Carolina
  - DM Clinical Research - Bellaire, Houston, Texas
  - DM Clinical Research - Tomball, Tomball, Texas